# CENTRAL SOUTH UNIVERSITY, XIANGYA SCHOOL OF NURSING YALE UNIVERSITY, YALE SCHOOL OF PUBLIC HEALTH

## **Qualitative Phone Interview – Consent Form for Participants**

Developing Efficient Intervention Technologies to Reduce Stigma-Related Stress, Mental Health Problems, and HIV Risk among Young Chinese MSM

Under the supervision of Xianhong Li, Ph.D., RN, & John Pachankis, Ph.D.

If available: Hello, I'm calling from the Yale School of Public Health and Central South University to talk about your experience in the Chinese ESTEEM iCBT study. The purpose of this research study is to test a type of online counseling intended to help young men who have sex with men (YMSM) in Hunan province China improve their sexual health and HIV risk behavior, as well as their ability to cope with symptoms of depression and anxiety. We want to thank you again for participating in our research and ask you a few final questions about your experience with the study, so that we can learn from you and improve it. These questions will take about 45-60 minutes to answer and will ask you to describe what worked well in the treatment delivery, if anything; what you liked and did not like about the study, if anything; and any suggestions you might have for how to make the treatment delivery better. You will receive 200 RMB for your participation.

Before we begin, I would like to go over some information about how we will use and protect the data that we collect from you today. It's very similar to what was outlined in the Chinese ESTEEM iCBT consent form, if you happen to remember that. But let's go over it briefly:

The information that you provide will be kept confidential. That is, your name will not be linked to the information you provide me except in the event that you report any intent to harm yourself or another person or child. In that case, I would have to waive confidentiality and take actions to protect you and/or others. Otherwise, the information you provide will be kept in a password-protected file on my computer, which no one will have access to other than myself and the Chinese ESTEEM iCBT research staff. Your therapist will not have access to this information. None of the information exchanged during this conversation will be made public or published in connection to your name. Some of the questions I will ask might bring up uncomfortable thoughts associated with the therapy sessions or may remind you of difficult past experiences you may have had. I'd like to get your consent to audio-record this interview so that we can later conduct analyses to learn from what you tell us today. I ask that you do not share your name or any other personally-identifying information, such as your address or friends' names, during this call, to help keep your information confidential. In the event that you accidently reveal any personally-identifiable information (e.g., your name) during the interview, this will be removed in the transcription. The audio recordings will be kept in a password-protected folder on my computer, which no one will have access to other than myself and the Chinese ESTEEM iCBT research staff. The audio recordings will be kept for three years after the study is completed, at which point they will be destroyed.

In addition to being regulated by applicable U.S. laws, the information you provide is protected by the General Data Protection Regulation, or 'GDPR', (EU) 2016/679 of the European Parliament and of the EU Council. The GDPR gives you certain rights with regard to your study data. You have the right to request access to, correction or erasure of, your study data. The project has support for the processing of personal data according to Article 6 (1) (a) of the EU Data Protection Regulation.

According to the EU Data Protection Regulation, you are entitled to obtain free information about all information about you that is handled within the study, and, if necessary, request that any errors be corrected. You may also

#### APPROVED BY THE YALE UNIVERSITY IRB 5/5/2022

request that information about you be deleted and that processing of your personal data be limited. If you want to request your information or request that your information be corrected, please contact Dr. Xianhong Li immediately at 86-731-82650264, or write to her at: 172 Tongzipo Road, Changsha, 410013, Hunan, China.

Taking part in this study is your choice. You can choose to take part, or you can choose not to take part in this study. You can also change your mind at any time. Whatever choice you make, you will not give up any legal rights or benefits. If you are interested in learning more about the study, please continue reading, or have someone read to you the rest of this document. Take as much time as you need before you make your decision. Ask the study staff questions about anything you do not understand. Once you understand the study, we will ask you if you wish to participate.

If you have any questions about the research study or experience a negative reaction that might have been caused by being in this study, please call Dr. Xianhong Li immediately at 86-731-82650264, or write to her at 172 Tongzipo Road, Changsha, 410013, Hunan, China

You should contact the Institutional Review Board at Xiangya School of Nursing of Central South University at 86-731-82650275 (86-18073185501) if you have questions about your rights as a research participant or to discuss research-related injuries.

Do you have any questions about what I just shared?

Do you consent to participate in this phone interview as part of the Chinese ESTEEM study? [If no, then thank them for their time and discontinue the phone call.]

Do you consent to have your responses audio-recorded as part of the Chinese ESTEEM study? [If no, then thank them for their time and discontinue the phone call.]

[BEGIN AUDIO RECORDING]

#### APPROVED BY THE YALE UNIVERSITY IRB 5/5/2022

### **Oualitative Phone Interview – Consent Form for Stakeholders**

Developing Efficient Intervention Technologies to Reduce Stigma-Related Stress, Mental Health Problems, and HIV Risk among Young Chinese MSM

Under the supervision of Xianhong Li, Ph.D., RN, & John Pachankis, Ph.D.

If available: Hello, I'm calling from the Yale School of Public Health and Central South University to talk about your experience or perspectives in the Chinese ESTEEM iCBT study. The purpose of this research study is to test a type of online counseling intended to help young men who have sex with men (YMSM) in Hunan province China improve their sexual health and HIV risk behavior, as well as their ability to cope with symptoms of depression and anxiety. We want to thank you again for participating in our interview and ask you a few questions about your perspectives with the study, so that we can learn from you and improve it. These questions will take about 45-60 minutes to answer and will ask you to describe what will work well in the treatment delivery, if anything; what you liked and did not like about the study, if anything; and any suggestions you might have for how to make the treatment delivery better. You will receive 200 RMB for your participation.

Before we begin, I would like to go over some information about how we will use and protect the data that we collect from you today. It's very similar to what was outlined in the Chinese ESTEEM iCBT consent form, if you happen to remember that. But let's go over it briefly:

The information that you provide will be kept confidential. That is, your name will not be linked to the information you provide me except in the event that you report any intent to harm yourself or another person or child. In that case, I would have to waive confidentiality and take actions to protect you and/or others. Otherwise, the information you provide will be kept in a password-protected file on my computer, which no one will have access to other than myself and the Chinese ESTEEM iCBT research staff. Your therapist will not have access to this information. None of the information exchanged during this conversation will be made public or published in connection to your name. Some of the questions I will ask might bring up uncomfortable thoughts associated with the therapy sessions or may remind you of difficult past experiences you may have had. I'd like to get your consent to audio-record this interview so that we can later conduct analyses to learn from what you tell us today. I ask that you do not share your name or any other personally-identifying information, such as your address or friends' names, during this call, to help keep your information confidential. In the event that you accidently reveal any personally-identifiable information (e.g., your name) during the interview, this will be removed in the transcription. The audio recordings will be kept in a password-protected folder on my computer, which no one will have access to other than myself and the Chinese ESTEEM iCBT research staff. The audio recordings will be kept for three years after the study is completed, at which point they will be destroyed.

In addition to being regulated by applicable U.S. laws, the information you provide is protected by the General Data Protection Regulation, or 'GDPR', (EU) 2016/679 of the European Parliament and of the EU Council. The GDPR gives you certain rights with regard to your study data. You have the right to request access to, correction or erasure of, your study data. The project has support for the processing of personal data according to Article 6 (1) (a) of the EU Data Protection Regulation.

According to the EU Data Protection Regulation, you are entitled to obtain free information about all information about you that is handled within the study, and, if necessary, request that any errors be corrected. You may also request that information about you be deleted and that processing of your personal data be limited. If you want to request your information or request that your information be corrected, please contact Dr. Xianhong Li immediately at 86-731-82650264, or write to her at: 172 Tongzipo Road, Changsha, 410013, Hunan, China.

#### APPROVED BY THE YALE UNIVERSITY IRB 5/5/2022

Taking part in this study is your choice. You can choose to take part, or you can choose not to take part in this study. You can also change your mind at any time. Whatever choice you make, you will not give up any legal rights or benefits. If you are interested in learning more about the study, please continue reading, or have someone read to you the rest of this document. Take as much time as you need before you make your decision. Ask the study staff questions about anything you do not understand. Once you understand the study, we will ask you if you wish to participate.

If you have any questions about the research study or experience a negative reaction that might have been caused by being in this study, please call Dr. Xianhong Li immediately at 86-731-82650264, or write to her at 172 Tongzipo Road, Changsha, 410013, Hunan, China

You should contact the Institutional Review Board at Xiangya School of Nursing of Central South University at 86-731-82650275 (86-18073185501) if you have questions about your rights as a research participant or to discuss research-related injuries.

Do you have any questions about what I just shared?

Do you consent to participate in this phone interview as part of the Chinese ESTEEM study? [If no, then thank them for their time and discontinue the phone call.]

Do you consent to have your responses audio-recorded as part of the Chinese ESTEEM study? [If no, then thank them for their time and discontinue the phone call.]

[BEGIN AUDIO RECORDING]